CLINICAL TRIAL: NCT00015548
Title: Comparative Effectiveness of Antipsychotic Medications in Patients With Alzheimer's Disease (CATIE Alzheimer's Disease Trial)
Brief Title: CATIE-Alzheimer's Disease Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH090001-05; N01 MH90001-AD; DSIR AT; N01MH90001 (NIH); N01MH090001 (NIH)
Record Dates: First submitted 2001-04-20; First posted 2001-04-23 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2009-02

CONDITIONS: Alzheimer's Disease
Keywords: antipsychotic treatment; Alzheimer's disease; agitation; dementia; psychosis; behavioral symptoms; hallucinations; delusions
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Dementia; Psychotic Disorders; Behavioral Symptoms; Hallucinations; Delusions | interventions — Olanzapine; Quetiapine Fumarate; Risperidone; Citalopram

INTERVENTIONS:
Drug: Olanzapine
Drug: Quetiapine
Drug: Risperidone
Drug: Citalopram

SUMMARY:
The CATIE Alzheimer's Disease Trial is part of the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Project. The study is for people with Alzheimer's disease who are having trouble with their thinking or behavior. In particular, this study is trying to find out the best treatment for people who have hallucinations (seeing or hearing things that aren't there), delusions (false beliefs), or agitation. The design of the trial helps to increase the chance that participants in the study receive a medication that helps them. The study uses three medications known as atypical antipsychotics (olanzapine, quetiapine, risperidone), which are the newest medications that are currently available for treating these problems. Participants may also receive an antidepressant (citalopram). The trial lasts for 36 weeks. Participants are given a thorough evaluation at no cost to ensure that this study is appropriate. In addition, the caregiver, family member, or friend who comes with the participant will be offered an educational program about Alzheimer's disease.

DETAILED DESCRIPTION:
There are four phases.

Phase I: In the initial treatment phase (Phase 1), patients will be randomized to one of the three atypical antipsychotics or placebo in the ratio 100:100:100:150 respectively. After two weeks, the investigator can move the patient to the next phase because of lack of efficacy or tolerability. At week 12, the investigator can decide whether the current medication is sufficiently optimal or it would be more beneficial to try another randomized medication.

Phase 2: Phase 2 starts when the patient is randomized to a second medication, i.e., olanzapine, quetiapine, risperidone, or citalopram. Patients will be randomized from an antipsychotic treatment to another antipsychotic treatment or citalopram in the ratio 3:3:2, or from placebo to an antipsychotic treatment or citalopram in the ratio 1:1:1:3 respectively. Therefore, 50% of patients who took placebo in Phase 1 will be randomized to an antipsychotic in Phase 2, and 50% will be randomized to citalopram in Phase 2. After the initial two weeks in Phase 2, the investigator can move the patient to the next phase, due to lack of efficacy or tolerability. After the patient has been on the Phase 2 study drug for approximately 12 weeks, the investigator can decide whether the current medication is sufficiently optimal or whether it would be more beneficial to try another randomized medication.

Phase 3: Phase 3 is randomized open-label treatment of one of the medications not previously received, i.e., olanzapine, quetiapine, risperidone, or citalopram. Treatment failures to the second treatment can be switched to a third open-label treatment. During Phase 3 patients will be maintained on their treatments openly and managed clinically until week 36.

If the investigator determines that the patient's response is not sufficiently optimal to the randomized open-label medication, then after the first two weeks of Phase 3, the investigator can prescribe another medication (of the investigator's choice) to the patient. If this occurs then patients are classed as being in the Open-Choice Phase.

Open-Choice Phase: The Open-Choice Phase can be entered at anytime during the 36-week study and directly from any of the three phases. There are four reasons a patient can enter the open choice phase:

* Withdrawal from Phase 1 or Phase 2 with the patient or surrogate decision-maker refusing to proceed to the next randomized phase;
* Withdrawal from Phase 3;
* Withdrawal from current study drug from any of the three previous phases due to antipsychotic medication no longer being required in the opinion of the investigator; or
* Withdrawal due to concomitant treatment with an exclusionary medication.

The Open-Choice Phase is designed to keep patients monitored in the trial for the 36-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Dementia of the Alzheimer's Type
* Ambulatory, Outpatients who have an informant living/visiting at least 8 hours/week over 3-4 days.
* Presence of delusions, hallucinations, agitation impacting functioning and requiring medication treatment
* Agitation or psychotic symptoms began after signs or symptoms of dementia

Exclusion (prospective participants must not:)

* Be benefiting from psychotropic medication, antidepressants or anticonvulsants
* Be diagnosed with schizophrenia, schizoaffective disorder, delusional disorder or mood disorder with psychotic features.
* Have severe or unstable medical illness requiring active treatment
* Have hypersensitivity or intolerance of any of the study medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2001-03; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Lon Schneider, MD, Principal Investigator — University of Southern California; Pierre Tariot, MD, Principal Investigator — University of Rochester
Locations (34):
- United States (34):
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - University of California, Irvine Medical Center, Irvine, California
  - University of Southern California Dept of Psychiatry& Behavioral Sciences, Los Angeles, California
  - University of California, Los Angeles, VA Medical Center, Los Angeles, California
  - University of California-San Diego, VA Medical Center, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Mental Health Advocates, Inc., Boca Raton, Florida
  - Berma Research Group, Hialeah, Florida
  - University of South Florida Suncoast Gerontology Center, Tampa, Florida
  - Palm Beach Neurology/Premiere Research Institute, West Palm Beach, Florida
  - Emory University - Wesley Woods Health Center, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Northwestern University Medical School, Chicago, Illinois
  - Southern Illinois School of Medicine, Springfield, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Millennium Psychiatric Associates, St Louis, Missouri
  - University of Medicine and Dentistry of New Jersey, Piscataway, New Jersey
  - University of Medicine and Dentistry of New Jersey-Stratford, Stratford, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Global Research and Consulting, Olean, New York
  - Monroe Community Hospital, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University Hospital Health Systems-Laurelwood Hospital, Willoughby, Ohio
  - VA Medical Center, Coatesville, Pennsylvania
  - Mental Illness Research Education and Clinical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Southwestern Vermont Medical Center- The Memory Clinic, Bennington, Vermont

REFERENCES:
- [Background] Schneider LS, Tariot PN, Lyketsos CG, Dagerman KS, Davis KL, Davis S, Hsiao JK, Jeste DV, Katz IR, Olin JT, Pollock BG, Rabins PV, Rosenheck RA, Small GW, Lebowitz B, Lieberman JA. National Institute of Mental Health Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE): Alzheimer disease trial methodology. Am J Geriatr Psychiatry. 2001 Fall;9(4):346-60. PMID 11739062
- [Background] Schneider LS, Ismail MS, Dagerman K, Davis S, Olin J, McManus D, Pfeiffer E, Ryan JM, Sultzer DL, Tariot PN. Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE): Alzheimer's disease trial. Schizophr Bull. 2003;29(1):57-72. doi: 10.1093/oxfordjournals.schbul.a006991. PMID 12908661
- [Result] Schneider LS, Tariot PN, Dagerman KS, Davis SM, Hsiao JK, Ismail MS, Lebowitz BD, Lyketsos CG, Ryan JM, Stroup TS, Sultzer DL, Weintraub D, Lieberman JA; CATIE-AD Study Group. Effectiveness of atypical antipsychotic drugs in patients with Alzheimer's disease. N Engl J Med. 2006 Oct 12;355(15):1525-38. doi: 10.1056/NEJMoa061240. PMID 17035647
- [Derived] Reeves S, Bertrand J, Uchida H, Yoshida K, Otani Y, Ozer M, Liu KY, Bramon E, Bies R, Pollock BG, Howard R. Towards safer risperidone prescribing in Alzheimer's disease. Br J Psychiatry. 2021 May;218(5):268-275. doi: 10.1192/bjp.2020.225. PMID 33176899
- [Derived] Nagata T, Shinagawa S, Yoshida K, Noda Y, Shigeta M, Mimura M, Nakajima S. Early Improvements of Individual Symptoms With Antipsychotics Predict Subsequent Treatment Response of Neuropsychiatric Symptoms in Alzheimer's Disease: A Re-Analysis of the CATIE-AD Study. J Clin Psychiatry. 2020 Feb 11;81(2):19m12961. doi: 10.4088/JCP.19m12961. PMID 32074412
- [Derived] Ozawa C, Roberts R, Yoshida K, Suzuki T, Lebowitz B, Reeves S, Howard R, Abe T, Mimura M, Uchida H. Placebo Effects in the Treatment of Noncognitive Symptoms of Alzheimer's Disease: Analysis of the CATIE-AD Data. J Clin Psychiatry. 2017 Nov/Dec;78(9):e1204-e1210. doi: 10.4088/JCP.17m11461. PMID 29045769
- [Derived] Yoshida K, Roberts R, Suzuki T, Lebowitz B, Reeves S, Howard R, Abe T, Mimura M, Uchida H. Lack of Early Improvement with Antipsychotics is a Marker for Subsequent Nonresponse in Behavioral and Psychological Symptoms of Dementia: Analysis of CATIE-AD Data. Am J Geriatr Psychiatry. 2017 Jul;25(7):708-716. doi: 10.1016/j.jagp.2017.01.016. Epub 2017 Jan 30. PMID 28215900
- [Derived] Miller EA, Schneider LS, Rosenheck RA. Predictors of nursing home admission among Alzheimer's disease patients with psychosis and/or agitation. Int Psychogeriatr. 2011 Feb;23(1):44-53. doi: 10.1017/S1041610210000244. Epub 2010 Mar 10. PMID 20214847
- [Derived] Zheng L, Mack WJ, Dagerman KS, Hsiao JK, Lebowitz BD, Lyketsos CG, Stroup TS, Sultzer DL, Tariot PN, Vigen C, Schneider LS. Metabolic changes associated with second-generation antipsychotic use in Alzheimer's disease patients: the CATIE-AD study. Am J Psychiatry. 2009 May;166(5):583-90. doi: 10.1176/appi.ajp.2008.08081218. Epub 2009 Apr 15. PMID 19369318
- [Derived] Sultzer DL, Davis SM, Tariot PN, Dagerman KS, Lebowitz BD, Lyketsos CG, Rosenheck RA, Hsiao JK, Lieberman JA, Schneider LS; CATIE-AD Study Group. Clinical symptom responses to atypical antipsychotic medications in Alzheimer's disease: phase 1 outcomes from the CATIE-AD effectiveness trial. Am J Psychiatry. 2008 Jul;165(7):844-54. doi: 10.1176/appi.ajp.2008.07111779. Epub 2008 Jun 2. PMID 18519523
- [Derived] Rosenheck RA, Leslie DL, Sindelar JL, Miller EA, Tariot PN, Dagerman KS, Davis SM, Lebowitz BD, Rabins P, Hsiao JK, Lieberman JA, Schneider LS; Clinical Antipsychotic Trial of Intervention Effectiveness-Alzheimer's Disease (CATIE-AD) investigators. Cost-benefit analysis of second-generation antipsychotics and placebo in a randomized trial of the treatment of psychosis and aggression in Alzheimer disease. Arch Gen Psychiatry. 2007 Nov;64(11):1259-68. doi: 10.1001/archpsyc.64.11.1259. PMID 17984395
- See also: More information about Alzheimer's Disease — http://www.alzheimers.org